CLINICAL TRIAL: NCT02716441
Title: Failure With Continuity and Its Relation to Rotator Cuff Repair Clinical Outcomes
Brief Title: Rotator Cuff Failure With Continuity
Status: Active, not recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Kathleen Derwin, PhD, Associate Staff, The Cleveland Clinic
Other Study IDs: 16-089
Record Dates: First submitted 2016-03-15; First posted 2016-03-23 (Estimated); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Rotator Cuff Tear
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- Radio-opaque Tissue Markers: Patients undergoing rotator cuff repair with implantation of radio-opaque tissue markers
  Interventions: Device: Radio-opaque Tissue Markers

INTERVENTIONS:
Device: Radio-opaque Tissue Markers — All participants will undergo implantation of radio-opaque tissue markers on their repaired rotator cuff at the time of surgery.

SUMMARY:
This proposal's objective is to challenge and expand the current definition of rotator cuff healing by investigating tendon retraction - broadly defined as medial translation of the repaired tendon away from the bone with or without a defect - as a common and clinically predictive structural outcome following rotator cuff repair. The investigators' central hypothesis is that failure with continuity is a common yet unrecognized structural phenomenon of rotator cuff healing that is significantly and meaningfully correlated with clinical outcomes. The investigators' approach is to characterize tendon retraction using an array of implanted radio-opaque markers, and investigate its relationship to pre-operative tissue quality (MRI), post-operative repair structural integrity (MRI) and clinical outcomes in a 125-patient prospective cohort study. These patients will complete (1) validated questionnaires and range of motion testing pre-operatively, (2) CT imaging at day of surgery, 3 weeks, 3 and 6 months, and 1, 2 and 5 years post-operatively, (3) MRI at 3 weeks, 3 and 6 months, and 1, 2 and 5 years post-operatively and (4) questionnaires, range of motion and strength testing at 3 and 6 months and 1, 2 and 5 years post-operatively.

DETAILED DESCRIPTION:
Currently, rotator cuff healing is defined as "intact", "attenuated", or "failed" based on the observation (or not) of a recurrent defect (i.e., a "gap") in the tendon using MRI or ultrasound imaging. The investigators' previous work has identified a new outcome, in which there is no detectable defect or "gap" in the repaired tendon, but the repaired tendon has undergone significant retraction. The investigators call this outcome "failure with continuity".

Current imaging methods are inadequate to determine the extent to which the repaired rotator cuff tendon has "failed with continuity". The investigators have developed an imaging technique to detect this phenomenon. Specifically, radio-opaque markers are sutured onto the repaired tendon. The distance between the tendon markers and the bone is measured from CT scans taken within 2 weeks of surgery, and compared to the distance measured at 3 and 6 months and 1, 2 and 5 years post-operatively. If the tendon retracts away from the bone during healing, this distance will increase over time. Healing of the tendon will also be monitored in the traditional manner by MRI scans at the same time points. The investigators will investigate the relationship between tendon retraction, MR imaging and clinical outcomes including shoulder strength and patient satisfaction.

The investigators expect to show that tendon retraction is common, occurs early post-operatively, with or without repair continuity as assessed by traditional imaging, and significantly correlates with clinical outcomes. The immediate and highly significant consequence of this finding would be a paradigm shift in the investigators' understanding of tendon repair healing, now incorporating the magnitude, timing and location of tendon retraction as well as the continuity of the repaired tissue. This information would yield a more precise understanding of rotator cuff tendon healing, allowing for advances in treatment strategies that improve surgical healing and clinical outcomes and result in more durable rotator cuff repairs over time.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, ages 18-75 having an acute or chronic 1-5 cm wide (A-P) full thickness tear of only the supraspinatus and/or infraspinatus tendons; partial thickness tears of subscapularis or teres minor not requiring repair are allowed.
* The tear must be fully reparable arthroscopically by a double row technique.
* Final determination of eligibility will be made at surgery when above inclusion criteria are confirmed.

Exclusion Criteria:

* Prior shoulder surgery (including rotator cuff repair)
* Symptomatic cervical spine disease
* A frozen shoulder-- defined as a loss of passive range of motion (ROM) of more than 20° in any plane compared to the contralateral shoulder,
* Glenohumeral arthritis grade 3 or 4-- defined as full thickness cartilage loss on MRI and confirmed at arthroscopy
* Worker's compensation cases
* Subscapularis tears of any size that require repair

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Study Population includes males and females between the ages of 18-75 who are undergoing arthroscopic rotator cuff repair surgery. Patients will be enrolled on a first come basis. No specific study demographic is necessary or desired.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in Tendon Retraction | Day of surgery and 1, 2 and 5 years following rotator cuff repair
  Medial translation of the repaired tendon away from the bone between the day of surgery and 1, 2 and 5 years following rotator cuff repair as measured by CT imaging of radio-opaque markers implanted on the tendon.

SECONDARY OUTCOMES:
Change in Shoulder Strength | Day of surgery and 1, 2 and 5 years following rotator cuff repair
  Isometric shoulder strength will be measured using a dynamometer.
Change in American Shoulder and Elbow Society (ASES) Score | Day of surgery and 1, 2 and 5 years following rotator cuff repair
  Patient reported outcome measure
Change in Pennsylvania Shoulder Score (PSS) | Day of surgery, and 1, 2 and 5 years following rotator cuff repair
  Patient reported outcome measure
Tendon Integrity | 1, 2 and 5 years following rotator cuff repair
  Traditional assessment of tendon repair integrity will be performed by MR imaging

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Derwin, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Main Campus, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No